CLINICAL TRIAL: NCT00625443
Title: A Phase 2, Parallel Group, Rollover Study of AKR-501 in Patients With Chronic Idiopathic Thrombocytopenic Purpura (ITP) Who Completed 28 Days of Study Treatment in Protocol 501-CL-003
Brief Title: Phase 2, Parallel Group, Rollover Study of AKR-501 in Patients With ChronicITP Who Completed 28 Days of Study Treatment in Protocol 501-CL-003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AKR-501-CL-004
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Results first posted 2018-03-16 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Idiopathic Thrombocytopenic Purpura
Keywords: Idiopathic Thrombocytopenic Purpura; ITP; Chronic Idiopathic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — avatrombopag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (double-blind) (Experimental)
  Interventions: Drug: Blinded (placebo)
- Avatrombopag tablets (open-label) (Experimental)
  Interventions: Drug: Open Label (Avatrombopag tablets)
- Avatrombopag tablets (double-blind) (Experimental)
  Interventions: Drug: Blinded (Avatrombopoag tablets)

INTERVENTIONS:
Drug: Blinded (placebo) — Placebo Orally, once daily administered under fasting conditions (at least 1 hr prior to or at least 2 hours after a meal or snack)
  Duration - 6 months
  Arms: Placebo (double-blind)
Drug: Open Label (Avatrombopag tablets) — Dose 10 mg
  Orally, once daily administered under fasting conditions (at least 1 hr prior to or at least 2 hours after a meal or snack)
  Duration - 6 months
  Other Names: AKR-501; E5501; YM477
  Arms: Avatrombopag tablets (open-label)
Drug: Blinded (Avatrombopoag tablets) — Dose: 2.5, 5, 10, or 20 mg
  Orally, once daily administered under fasting conditions (at least 1 hr prior to or at least 2 hours after a meal or snack)
  Duration - 6 months
  Other Names: AKR-501; E5501; YM477
  Arms: Avatrombopag tablets (double-blind)

SUMMARY:
The purpose of this study is to determine the safety and efficacy of AKR-501 (avatrombopag) administered in participants with chronic Idiopathic Thrombocytopenic Purpura (ITP) who were enrolled into and completed 28 days of study treatment in Protocol 501-CL-003 (NCT00441090).

DETAILED DESCRIPTION:
Participants eligible to enroll into this rollover protocol will begin study treatment within 2-5 days of their Day 28 study termination visit in Protocol 501-CL-003 (NCT00441090). Participants who met the primary efficacy response criterion in Protocol 501-CL-003 will continue receiving the same study treatment to which they were assigned in the previous protocol in a double-blinded manner, these being one of the following 5 treatments:

* avatrombopag 2.5 mg daily
* avatrombopag 5 mg daily
* avatrombopag 10 mg daily
* avatrombopag 20 mg daily
* placebo

Participants who did not meet the primary efficacy response criterion in Protocol 501-CL-003 who otherwise meet the eligibility criteria for this rollover protocol will be offered open label avatrombopag 10 mg daily.

This is a parallel group, rollover study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who completed 28 days of study treatment in Protocol 501-CL-003.
2. No significant safety or tolerability concerns from the patient's participation of Protocol 501-CL-003 as determined by the Investigator.
3. Received medical monitor approval for enrollment into this study.
4. Patients receiving maintenance corticosteroids may be enrolled, as long as the corticosteroids have been administered at a stable dose and the Investigator does not foresee the need to change the steroid dose during study participation. Patients should remain on this stable corticosteroid dose during study participation.
5. Women of child-bearing potential must have a negative serum pregnancy test at the Day 28 assessment in Protocol 501-CL-003. (Childbearing potential is defined as any woman who has not been surgically sterilized and is pre-menopausal or peri-menopausal i.e., any menstrual flow within 12 months of Screening Visit A for Protocol 501-CL-003).
6. Women of child-bearing potential must agree to practice a medically approved form of contraception (one of the following must be used: condoms (male or female) with a spermicidal agent, diaphragm or cervical cap with a spermicidal agent, IUD,hormonal contraception, abstinence).
7. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Women who are pregnant and/or lactating.
2. Use of the following drugs or treatments:

   * Rituximab
   * Azathioprine, Cyclosporine A, or other immunosuppressant therapy
   * Aspirin, Aspirin-containing compounds, Salicylates,Anticoagulants, Non-steroidal anti-inflammatory drugs(NSAIDs)(including Cyclooxygenase-2 [COX-2] specific NSAIDs), clopidogrel; ticlopidine; and any drugs that affect platelet function.
   * Danazol
   * Rh0(D) immune globulin (WinRho®) or intravenous immunoglobulin (IVIG).
3. Inability to comply with protocol requirements or give informed consent, as determined by the Investigator.

For more information regarding inclusion/exclusion criteria, please see record for AKR 501-CL-003 Protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-05; Primary Completion 2009-06 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Ran Ho, MD, Study Director — Eisai Inc.
Locations (12):
- United States (12):
  - Pacific Cancer Medical Center, Inc, Anaheim, California
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Davis, Posteraro and Wasser, MDs, LLP, Manchester, Connecticut
  - Florida Cancer Institute, New Port Richey, Florida
  - John H. Stroger, Jr. Hospital of Cook County, Div. of Hematology and Oncology, Chicago, Illinois
  - Cancer Care Center, Inc., New Albany, Indiana
  - Capitol Comprehensive Cancer Care Clinic, Jefferson City, Missouri
  - Kansas City Cancer Center, LLC, Kansas City, Missouri
  - Mount Sinai Medical Center, New York, New York
  - New York Presbyterian Hospital, Weill Medical College of Cornell University, New York, New York
  - Emerywood Oncology and Hematology, High Point, North Carolina
  - Mid Ohio Oncology/Hematology, Inc., dba The Mark H. Zangmeister Center, Columbus, Ohio

REFERENCES:
- [Derived] Bussel JB, Kuter DJ, Aledort LM, Kessler CM, Cuker A, Pendergrass KB, Tang S, McIntosh J. A randomized trial of avatrombopag, an investigational thrombopoietin-receptor agonist, in persistent and chronic immune thrombocytopenia. Blood. 2014 Jun 19;123(25):3887-94. doi: 10.1182/blood-2013-07-514398. Epub 2014 May 6. PMID 24802775

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After Protocol Amendment 4, this study implemented a flexible dose regimen and was considered to have an open-label, uncontrolled, single-arm design. Due to these limitations in study design, a single grouping method with 3 subgroups was implemented for reporting participant disposition.
Groups:
- Lower 1/3 Avatromboopag Dose Group: Participants in this group took less than 8.85 mg avatrombopag orally once daily under fasting conditions (at least 1 hour before and 2 hours after a meal or snack). Grouping of avatrombopag dose into lower 1/3, middle 1/3, and upper 1/3 was based on the average daily dose received during the combined active treatment periods of studies 501-CL-003 and 501-CL-004.
- Middle 1/3 Avatrombopag Dose Group: Participants in this group took greater than or equal to 8.85 mg avatrombopag to less than 13.5 mg avatrombopag orally once daily under fasting conditions (at least 1 hour before and 2 hours after a meal or snack). Grouping of avatrombopag dose into lower 1/3, middle 1/3, and upper 1/3 was based on the average daily dose received during the combined active treatment periods of studies 501-CL-003 and 501-CL-004.
- Upper 1/3 Avatrombopag Dose Group: Participants in this group took greater than or equal to 13.5 mg avatrombopag orally once daily under fasting conditions (at least 1 hour before and 2 hours after a meal or snack). Grouping of avatrombopag dose into lower 1/3, middle 1/3, and upper 1/3 was based on the average daily dose received during the combined active treatment periods of studies 501-CL-003 and 501-CL-004.
Period: Overall Study
Arm/Group | Lower 1/3 Avatromboopag Dose Group | Middle 1/3 Avatrombopag Dose Group | Upper 1/3 Avatrombopag Dose Group
Started | 12 | 26 | 15
Completed | 10 | 15 | 10
Not Completed | 2 | 11 | 5
Not completed — Adverse Event | 1 | 4 | 0
Not completed — Non-compliance with protocol | 0 | 1 | 0
Not completed — Platelet count increase >=500,000/mm3 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2
Not completed — Physician Decision | 0 | 4 | 2
Not completed — Other | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who completed 501-CL-003 and received study drug in 501-CL-004, except baseline values and ITP-directed medications taken during the 2-week period before the first dose of avatrombopag in 501-CL-004. Data was summarized using the observed case (OC) method.
Groups:
- Lower 1/3 Avatrombopag Dose Group: Participants in this group took less than 8.85 mg avatrombopag orally once daily under fasting conditions (at least 1 hour before and 2 hours after a meal or snack). Grouping of avatrombopag dose into lower 1/3, middle 1/3, and upper 1/3 was based on the average daily dose received during the combined active treatment periods of studies 501-CL-003 and 501-CL-004.
- Total: Total of all reporting groups
Arm/Group | Lower 1/3 Avatrombopag Dose Group | Middle 1/3 Avatrombopag Dose Group | Upper 1/3 Avatrombopag Dose Group | Total
Number analyzed (Participants) | 12 | 26 | 15 | 53
Age, Continuous [Geometric Mean (Standard Deviation); unit: Years] | 44.7 (21.09) | 52.5 (18.44) | 50.4 (15.65) | 50.1 (18.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 20 | 11 | 38
  Male | 5 | 6 | 4 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: A TEAE was defined as 1) the AE started on or after the date of first dose of study drug up to and including 30 days after the last dose of study drug, or 2) the AE started before the first dose of study drug but worsened in severity on or after the date of first dose of study drug up to and including 3 days after the last dose of study drug. For participants having a tapering period of study drug, the last dose day is the last day of study drug during the tapering period. Related AEs included those whose relationship was categorized as possible or probably by the investigator. Dose interruption includes dose decreased, dose previously stopped, permanently stopped, or temporarily stopped. The safety population was divided into three subgroups based on the mean daily dose of active study drug taken; lower 1/3 (less than 8.85 mg avatrombopag), middle 1/3 (greater than or equal to 8.85 mg but less than 13.5 mg avatrombopag), and upper 1/3 (greater than or equal to 13.5 mg avatrombopag).
Time Frame: Day 1 through Month 6 while receiving treatment and at Month 7 after discontinuation of treatment.
Population: Safety population included all participants who received at least one dose of study drug and had at least one post-treatment safety assessment. The term "post-treatment" refers to any assessment timepoint after the participant received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Lower 1/3 Avatrombopag Dose Group | Middle 1/3 Avatrombopag Dose Group | Upper 1/3 Avatrombopag Dose Group
Number analyzed (Participants) | 12 | 26 | 15
Participants
  TEAEs | 12 | 24 | 14
  Severe (Grade 3-4) TEAEs | 4 | 7 | 6
  Treatment-related TEAEs | 5 | 15 | 7
  Serious TEAEs | 2 | 4 | 3
  Serious treatment-related TEAEs | 1 | 2 | 0
  Withdrawal of study drug due to TEAE | 2 | 4 | 0
  Dose interruption due to TEAE | 2 | 3 | 2
  Deaths | 0 | 0 | 0

2. Primary Outcome: Incidence of Severe (Grade 3 or 4) TEAEs
Description: A TEAE was defined as 1) the AE started on or after the date of first dose of study drug up to and including 30 days after the last dose of drug, or 2) the AE started before the first dose of study drug but worsened in severity on or after the date of first dose of study drug up to and including 3 days after the last dose of study drug. For participants having a tapering period of study drug, the last dose day is the last day of study drug during the tapering period. The safety population was divided into three subgroups based on the mean daily dose of active study drug taken; lower 1/3 (less than 8.85 mg avatrombopag), middle 1/3 (greater than or equal to 8.85 mg but less than 13.5 mg avatrombopag), and upper 1/3 (greater than or equal to 13.5 mg avatrombopag).
Time Frame: Day 1 through Month 6 while receiving treatment and at Month 7 after discontinuation of treatment.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lower 1/3 Avatrombopag Dose Group | Middle 1/3 Avatrombopag Dose Group | Upper 1/3 Avatrombopag Dose Group
Number analyzed (Participants) | 12 | 26 | 15
Participants
  Thrombocytopenia | 1 | 2 | 4
  Splenomegaly | 0 | 0 | 1
  Haemorrhagic diathesis | 0 | 1 | 0
  Idiopathic thrombocytopenic purpura | 1 | 0 | 0
  Leukocytosis | 0 | 1 | 0
  Mitral valve incompetence | 0 | 0 | 1
  Diarrhoea | 0 | 0 | 1
  Vomiting | 0 | 0 | 1
  Fatigue | 2 | 0 | 0
  Oedema peripheral | 1 | 0 | 0
  Asthenia | 1 | 0 | 0
  Chest pain | 0 | 0 | 1
  Pyrexia | 0 | 0 | 1
  Platelet count increased | 2 | 1 | 0
  Platelet count decreased | 0 | 2 | 0
  Alanine aminotransferase increased | 0 | 0 | 1
  Aspartate aminotransferase increased | 0 | 0 | 1
  Hyperuricaemia | 1 | 0 | 0
  Back pain | 1 | 0 | 0
  Dizziness | 1 | 0 | 0
  Hypoaesthesia | 0 | 0 | 1
  Cerebrovascular accident | 0 | 0 | 1
  Haemorrhage intercranial | 0 | 1 | 0
  Epistaxis | 1 | 0 | 0
  Hypotension | 1 | 0 | 0
  Pelvic venous thrombosis | 0 | 1 | 0

3. Primary Outcome: Incidence of Drug-Related TEAEs
Description: Drug-related TEAEs included those whose relationship was categorized as possible or probably by the investigator. A TEAE was defined as 1) the AE started on or after the date of first dose of study drug up to and including 30 days after the last dose of drug, or 2) the AE started before the first dose of study drug but worsened in severity on or after the date of first dose of study drug up to and including 3 days after the last dose of study drug. For participants having a tapering period of study drug, the last dose day is the last day of study drug during the tapering period. The safety population was divided into three subgroups based on the mean daily dose of active study drug taken; lower 1/3 (less than 8.85 mg avatrombopag), middle 1/3 (greater than or equal to 8.85 mg but less than 13.5 mg avatrombopag), and upper 1/3 (greater than or equal to 13.5 mg avatrombopag).
Time Frame: Day 1 through Month 6 while receiving treatment and at Month 7 after discontinuation of treatment.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lower 1/3 Avatrombopag Dose Group | Middle 1/3 Avatrombopag Dose Group | Upper 1/3 Avatrombopag Dose Group
Number analyzed (Participants) | 12 | 26 | 15
Participants
  Thrombocytopenia | 1 | 2 | 0
  Splenomegaly | 0 | 1 | 1
  Anaemia | 0 | 1 | 0
  Leukocytosis | 0 | 1 | 0
  Vision blurred | 0 | 1 | 0
  Visual disturbance | 0 | 1 | 0
  Nausea | 0 | 0 | 2
  Abdominal pain upper | 0 | 0 | 1
  Diarrhoea | 0 | 1 | 0
  Vomiting | 0 | 0 | 1
  Fatigue | 2 | 4 | 1
  Oedema peripheral | 0 | 1 | 0
  Platelet count increased | 2 | 2 | 0
  Platelet count decreased | 0 | 2 | 0
  Alanine aminotransferase increased | 0 | 1 | 0
  Hyperlipidaemia | 2 | 1 | 0
  Decreased appetite | 0 | 0 | 1
  Arthralgia | 0 | 1 | 1
  Back pain | 0 | 0 | 2
  Pain in extremity | 0 | 2 | 0
  Arthropathy | 0 | 1 | 0
  Muscular weakness | 0 | 0 | 1
  Headache | 2 | 1 | 1
  Dizziness | 1 | 1 | 1
  Hypoaesthesia | 0 | 0 | 1
  Mood swings | 1 | 0 | 0
  Haematuria | 0 | 1 | 0
  Menorrhagia | 1 | 0 | 0
  Dyspnoea | 1 | 1 | 0
  Epistaxis | 1 | 0 | 1
  Nasal congestion | 0 | 0 | 1
  Rash | 0 | 1 | 0

4. Secondary Outcome: Median Platelet Counts at Selected Analysis Timepoints
Description: Platelet count (PC) was measured from blood draws. Based on avatrombopag response in study 501-CL-003, participants were divided into two subgroups; 1) "Responders", participants who met the primary efficacy response; pretreatment PC was less than 30,000/mm^3 and increased to greater than or equal to 50,000/mm^3 after treatment with avatrombopag, and for participants on steroids, pretreatment PC was greater than or equal to 30,000/mm3 but less than 50,000/mm^3 and increased to a PC greater than or equal to 20,000/mm^3 above their pretreatment values and 2) "Nonresponders", participants who did not meet the primary efficacy response and those who were in the placebo arm. Open-label dose escalation of avatrombopag, as well as reductions in ITP-directed concomitant therapy (e.g. steroids) was allowed for all participants. During the periods of avatrombopag dose escalation and/or ITP-directed concomitant medication reduction, platelet sampling was done weekly.
Time Frame: Day 1, Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, and Follow-up Weeks (after last dose of study drug in this study) 1, 2, 3, 4
Population: Full analysis set (FAS) included all participants who completed 501-CL-003 and received study drug in the current study, except baseline values and ITP-directed medications taken during the 2-week period before the first dose of avatrombopag in the current study. Data was summarized using the observed case (OC) method.
Measure: Median (Full Range); unit: Platelets x 1000/mm^3
Groups:
- Responders: Participants continued on their previous blinded dose in study 501-CL-003 at entry into this study. These blinded doses were: avatrombopag 2.5 mg, 5 mg, 10 mg, and 20 mg. The maximum possible escalated dose was a total dose of assigned double-blind avatrombopag plus an additional 20 mg/day open-label avatrombopag. Grouping Method B of dividing participants into Responders and Non-Responders was based on both treatment received and Day 28 platelet response to study drug in study 501-CL-004.
- Nonresponders: Participants began treatment with open-label 10 mg avatrombopag daily. The maximum possible escalated dose was 40 mg/day open-label. Grouping Method B of dividing participants into Responders and Non-Responders was based on both treatment received and Day 28 platelet response to study drug in study 501-CL-004.
Arm/Group | Responders | Nonresponders
Number analyzed (Participants) | 25 | 28
Platelets x 1000/mm^3
  Day 1 | 55.0 [7 to 316] | 23.5 [8 to 240]
  Week 2: number analyzed (Participants) | 22 | 28
  Week 2 | 126.0 [39 to 855] | 54.5 [5 to 1207]
  Week 4: number analyzed (Participants) | 24 | 27
  Week 4 | 113.0 [8 to 489] | 38.0 [6 to 383]
  Week 6: number analyzed (Participants) | 23 | 26
  Week 6 | 104.0 [18 to 880] | 47.0 [10 to 731]
  Week 8: number analyzed (Participants) | 21 | 26
  Week 8 | 137.0 [13 to 571] | 45.5 [3 to 263]
  Week 10: number analyzed (Participants) | 6 | 16
  Week 10 | 85.5 [32 to 179] | 72.0 [9 to 702]
  Week 12: number analyzed (Participants) | 14 | 20
  Week 12 | 88.0 [4 to 293] | 72.0 [2 to 557]
  Week 14: number analyzed (Participants) | 10 | 12
  Week 14 | 84.0 [29 to 296] | 77.5 [9 to 368]
  Week 16: number analyzed (Participants) | 11 | 17
  Week 16 | 143.0 [45 to 395] | 46.0 [3 to 273]
  Week 18: number analyzed (Participants) | 17 | 19
  Week 18 | 119.0 [28 to 303] | 78.0 [17 to 382]
  Week 20: number analyzed (Participants) | 10 | 12
  Week 20 | 92.0 [39 to 322] | 68.0 [18 to 481]
  Week 22: number analyzed (Participants) | 16 | 16
  Week 22 | 109.0 [26 to 354] | 78.5 [14 to 502]
  Week 24: number analyzed (Participants) | 21 | 17
  Week 24 | 154.0 [28 to 335] | 66.0 [19 to 368]
  Follow-up Week 1: number analyzed (Participants) | 11 | 11
  Follow-up Week 1 | 59.0 [8 to 495] | 40.0 [23 to 365]
  Follow-up Week 2: number analyzed (Participants) | 10 | 12
  Follow-up Week 2 | 25.0 [6 to 86] | 22.0 [8 to 426]
  Follow-up Week 3: number analyzed (Participants) | 12 | 9
  Follow-up Week 3 | 27.0 [3 to 380] | 36.0 [14 to 791]
  Follow-up Week 4: number analyzed (Participants) | 13 | 15
  Follow-up Week 4 | 35.0 [15 to 331] | 28.0 [1 to 881]

5. Secondary Outcome: Percentage of Participants Who Achieved a Platelet Count of 100,000/mm^3 or Higher by Response Status and Selected Study Visit
Description: Platelet count (PC) was measured from blood draws. Based on avatrombopag response in study 501-CL-003, participants were divided into two subgroups; 1) "Responders", participants who met the primary efficacy response; pretreatment PC was less than 30,000/mm^3 and increased to greater than or equal to 50,000/mm^3 after treatment with avatrombopag, and for participants on steroids, pretreatment PC was greater than or equal to 30,000/mm^3 but less than 50,000/mm^3 and increased to a PC greater than or equal to 20,000/mm^3 above their pretreatment values and 2) "Nonresponders", participants who did not meet the primary efficacy response and those who were in the placebo arm. Open-label dose escalation of avatrombopag, as well as reductions in ITP-directed concomitant therapy (e.g. steroids) was allowed for all participants. During the periods of avatrombopag dose escalation and/or ITP-directed concomitant medication reduction, platelet sampling was done weekly.
Time Frame: Baseline (last PC before first dose of study drug in previous study), Weeks 2, 4, 8, 12, 16, 20, 24, and Follow-up Weeks (after last dose of study drug in this study) 1, 2, 3, 4
Population: FAS. Data was summarized using the OC method.
Measure: Number; unit: Percentage of participants
Arm/Group | Responders | Nonresponders
Number analyzed (Participants) | 25 | 28
Percentage of participants
  Week 2 | 59.1 | 25.0
  Week 4 | 58.3 | 18.5
  Week 8 | 52.4 | 15.4
  Week 12 | 42.9 | 35.0
  Week 16 | 63.6 | 17.6
  Week 20 | 40.0 | 25.0
  Week 24 | 71.4 | 35.3
  Follow up Week 1 | 18.2 | 27.3
  Follow up Week 2 | 0 | 33.3
  Follow up Week 3 | 25.0 | 11.1
  Follow up Week 4 | 23.1 | 13.3

6. Secondary Outcome: Percentage of Participants Who Maintained a Platelet Count of 100,000/mm^3 or Higher by Response Status
Description: as for outcome 5
Time Frame: as for outcome 5
Population: FAS. Data was summarized using the OC method.
Measure: Number; unit: Percentage of participants
Arm/Group | Responders | Nonresponders
Number analyzed (Participants) | 25 | 28
Percentage of participants | 32.0 | 0

7. Secondary Outcome: Percentage of Participants Who Achieved Response-Level Platelet Count by Selected Study Visit
Description: as for outcome 5
Time Frame: as for outcome 5
Population: FAS. Data was summarized using the OC method.
Measure: Number; unit: Percentage of participants
Groups:
- Responders: Participants continued on their previous blinded dose study 501-CL-003 at entry into this study. These blinded doses were: avatrombopag 2.5 mg, 5 mg, 10 mg, and 20 mg. The maximum possible escalated dose was a total dose of assigned double-blind avatrombopag plus an additional 20 mg/day open-label avatrombopag. Grouping Method B of dividing participants into Responders and Non-Responders was based on both treatment received and Day 28 platelet response to study drug in study 501-CL-004.
Arm/Group | Responders | Nonresponders
Number analyzed (Participants) | 25 | 28
Percentage of participants
  Week 2 | 86.4 | 53.6
  Week 4 | 79.2 | 44.4
  Week 8 | 90.5 | 46.2
  Week 12 | 85.7 | 65.0
  Week 16 | 81.8 | 47.1
  Week 20 | 90.0 | 66.7
  Week 24 | 81.0 | 70.6
  Follow up Week 1 | 54.5 | 45.5
  Follow up Week 2 | 10.0 | 33.3
  Follow up Week 3 | 41.7 | 44.4
  Follow up Week 4 | 38.5 | 33.3

8. Secondary Outcome: Percentage of Participants Who Maintained Response-Level Platelet Count
Description: as for outcome 5
Time Frame: as for outcome 5
Population: FAS. Data was summarized using the OC method.
Measure: Number; unit: Percentage of participants
Arm/Group | Responders | Nonresponders
Number analyzed (Participants) | 25 | 28
Percentage of participants | 56.0 | 0

9. Secondary Outcome: Percentage of Participants Who Achieved a Durable, Transient, or Overall Platelet Response
Description: as for outcome 5
Time Frame: as for outcome 5
Population: FAS. Data was summarized using the OC method.
Measure: Number; unit: Percentage of participants
Arm/Group | Responders | Nonresponders
Number analyzed (Participants) | 25 | 28
Percentage of participants
  Durable Platelet Response | 72.0 | 35.7
  Transient Platelet Response | 16.0 | 28.6
  Overall Response | 88.0 | 64.3

10. Secondary Outcome: Number of Participants With Changes in Concomitant Steroid Use
Description: A participant who used steroids at study entry was considered to have permanently discontinued steroid use if they had no steroid use during the last 8 weeks of the study Treatment Period. A participant who used steroids at study entry was considered to have decreased concomitant steroid medication by at least 50% if they permanently discontinued steroids, or in no dose of steroid was higher than 50% of their baseline steroid dose during the last 8 weeks of the study Treatment Period.
Time Frame: Day 1 through last 8 weeks of the Treatment Period
Population: FAS. Data was summarized using the OC method. Only those participants who had data available at both Baseline and post-Baseline were analyzed.
Measure: Number; unit: Number of participants
Arm/Group | Responders | Nonresponders
Number analyzed (Participants) | 24 | 24
Number of participants
  Permanently Discontinued: number analyzed (Participants) | 12 | 12
  Permanently Discontinued | 4 | 4
  Decreased by greater than or equal to 50%: number analyzed (Participants) | 12 | 12
  Decreased by greater than or equal to 50% | 7 | 6

ADVERSE EVENTS:
Time Frame: Approximately 7 months.
Description: Treatment-emergent adverse events and treatment-emergent serious adverse events were reported. Safety population included all participants who received at least one dose of study drug and had at least one post-treatment safety assessment. The term "post-treatment" refers to any assessment timepoint after the participant received at least one dose of study drug.
Groups:
- Lower 1/3 Avatrombopag Dose Group: Participants in this group took less than 8.85 mg avatrombopag orally once daily under fasting conditions (at least 1 hour before and 2 hours after a meal or snack). Grouping Method A of avatrombopag dose into lower 1/3, middle 1/3, and upper 1/3 was based on the average daily dose received during the combined active treatment periods of studies 501-CL-003 and 501-CL-004.
- Middle 1/3 Avatrombopag Dose Group: Participants in this group took greater than or equal to 8.85 mg avatrombopag to less than 13.5 mg avatrombopag orally once daily under fasting conditions (at least 1 hour before and 2 hours after a meal or snack). Grouping Method A of avatrombopag dose into lower 1/3, middle 1/3, and upper 1/3 was based on the average daily dose received during the combined active treatment periods of studies 501-CL-003 and 501-CL-004.
- Upper 1/3 Avatrombopag Dose Group: Participants in this group took greater than or equal to 13.5 mg avatrombopag orally once daily under fasting conditions (at least 1 hour before and 2 hours after a meal or snack). Grouping Method A of avatrombopag dose into lower 1/3, middle 1/3, and upper 1/3 was based on the average daily dose received during the combined active treatment periods of studies 501-CL-003 and 501-CL-004.
Arm/Group | Lower 1/3 Avatrombopag Dose Group | Middle 1/3 Avatrombopag Dose Group | Upper 1/3 Avatrombopag Dose Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/26 | 0/15
Serious Adverse Events (participants affected / at risk) | 2/12 | 4/26 | 3/15
Other Adverse Events (participants affected / at risk) | 12/12 | 24/26 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lower 1/3 Avatrombopag Dose Group (N=12) | Middle 1/3 Avatrombopag Dose Group (N=26) | Upper 1/3 Avatrombopag Dose Group (N=15)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 2
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0
Pelvic venous thrombosis (Vascular disorders) | 0 | 1 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lower 1/3 Avatrombopag Dose Group (N=12) | Middle 1/3 Avatrombopag Dose Group (N=26) | Upper 1/3 Avatrombopag Dose Group (N=15)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3 | 4
Gingival bleeding (Gastrointestinal disorders) | 1 | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 1 | 3
Vomiting (Gastrointestinal disorders) | 0 | 2 | 2
Constipation (Gastrointestinal disorders) | 0 | 3 | 0
Fatigue (General disorders) | 5 | 4 | 4
Oedema peripheral (General disorders) | 1 | 2 | 3
Oedema (General disorders) | 1 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 1
Nasopharyngitis (Infections and infestations) | 2 | 1 | 0
Platelet count increased (Investigations) | 2 | 2 | 0
Platelet count decreased (Investigations) | 0 | 3 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Headache (Nervous system disorders) | 2 | 7 | 3
Dizziness (Nervous system disorders) | 1 | 1 | 2
Insomnia (Psychiatric disorders) | 1 | 2 | 1
Haematuria (Renal and urinary disorders) | 0 | 2 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 3 | 1 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 3 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other